CLINICAL TRIAL: NCT04319705
Title: Effects of Azithromycin Treatment on Anti-viral Immunity in Patients With Asthma and COPD - A Randomized Double-blind, Placebo-controlled Trial
Brief Title: Anti-viral Effects of Azithromycin in Patients With Asthma and COPD
Acronym: AZIMUNE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Lund University (Other); University of Copenhagen (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Celeste Porsbjerg, Professor, MD, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0052256
Record Dates: First submitted 2020-03-12; First posted 2020-03-24 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Asthma; COPD; Exacerbation Copd; Asthma; Eosinophilic; Bronchial Diseases; Lung Diseases, Obstructive; Lung Diseases; Immune System Diseases
Keywords: Eosinophil; Smoking; COPD; Asthma; Rhinovirus; Azithromycin; Inflammation; Microbiome
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Pulmonary Eosinophilia; Bronchial Diseases; Lung Diseases, Obstructive; Lung Diseases; Immune System Diseases; Smoking; Inflammation | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin (Experimental): Azithromycin, 500mg capsule, 3 times per week, during a 12-week period, administered orally
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Apart from the active substance, the placebo is otherwise identical to IMP, capsule, 3 times per week, during a 12-week period, administered orally
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Azithromycin — Azithromycin, 500mg, 3 times per week, 12-week treatment period, administered orally
  Arms: Azithromycin
Drug: Placebo oral tablet — capsule containing placebo, 3 times per week, 12-week treatment period, administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the anti-viral effects of low-dose AZM treatment in patients with asthma and COPD with an exacerbation history.

The investigators expect that long-term treatment with low dose AZM modulates the immune response to viral infections, with an increased interferon release, in patients with asthma and COPD with an exacerbation history. In addition, the investigators expect a decrease in inflammatory cells and mediators, and changes in bacteria, measured in samples from the lungs.

Half of the participants will receive azithromycin on top of their regular asthma/COPD treatment, while the other half will receive placebo on top of their regular asthma/COPD treatment.

DETAILED DESCRIPTION:
Asthma and COPD are responsible for considerable global morbidity and healthcare costs, primarily driven by exacerbations, i.e. acute flare-ups. Hence there is a clear need for better interventions preventing exacerbations. A majority of exacerbations are driven by infections, and in particular viral infections. Importantly, the anti-viral defense in asthma and COPD seems compromised, with a relative inability to combat infections, but also a disproportionate inflammatory response to infections, i.e. an increased immunoreactivity involving release of epithelial 'alarmins', such as IL-33 and thymic stromal lymphopoietin (TSLP).

Long-term low dose macrolides have been shown to reduce exacerbations in both diseases and are increasingly used clinically, but the mechanism of action is unknown. Macrolides have anti-viral properties in vitro, however their anti-viral properties have not been established in patients with asthma and COPD during exacerbations.

The purpose of this study is to investigate the anti-viral and anti-inflammatory effects in the airways, as well as the effects of azithromycin on the lung microbiome. In order to study these effects, the key endpoints in this trial will need to be obtained from bronchoscopic sampling of bronchial brushes, bronchial biopsies and BAL. But performing bronchoscopies during acute exacerbations, when patients are infected with respiratory viruses, is difficult in view of safety. Therefore, this study on in vitro rhinovirus responses of human bronchial epithelial cells before and after in vivo treatment with macrolides represents a novel model to study treatment effects on immunoreactivity during exacerbations.

The investigators hypothesize that long-term treatment with low dose AZM modulates the immune response to viral infections, with an increased interferon release, in patients with asthma and COPD with an exacerbation history.

The investigators also speculate that AZM treatment leads to a decreased release of the epithelial alarmins (e.g. IL-33 and TSLP) in response to viral infection, in patients with asthma and COPD with an exacerbation history.

Furthermore, treatment effects of low dose AZM on functional and compositional changes of bacterial communities of the respiratory- and gastrointestinal tract, and their association with changes in immunoreactivity will be studied.

This trial offers the opportunity to study potential biomarkers and surrogate endpoints, but also to identify the anti-inflammatory effects of azithromycin on a mechanistic level.

This study is a randomized, double-blind, placebo-controlled trial. It includes a enrolment period of maximum 4 weeks, with a bronchoscopy before and after 12 weeks of treatment (500mg azithromycin or placebo, 3 times per week).

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients (n=40)

  1. Diagnosis of asthma according to GINA, with confirmed variable airflow obstruction at screening visit or previously.
  2. Age ≥ 18 through 75 years.
  3. A postbronchodilator FEV1 ≥ 50% predicted
  4. Maintenance treatment with ICS and ≥ 1 second controller (LABA, LAMA, LTRA or Xanthines) for at least three months prior to Visit 1.
  5. Non-smokers (<10 packyears, quit >6 months).
  6. ≥ 1 Systemic steroid treated exacerbation in the past one year despite maintenance treatment with inhaled corticosteroids.
  7. Eosinophilic (n=20, blood eosinophils ≥ 0.200x109/L) and non-eosinophilic (n=20, blood eosinophils <0.200x109/L) phenotypes.
* COPD patients (n=40)

  1. Diagnosis of COPD according to GOLD
  2. Age ≥ 45 through 75 years.
  3. ≥ 10 packyears smoking history (current or ex-smokers).
  4. A postbronchodilator FEV1 ≥ 30% predicted.
  5. Maintenance treatment with long-acting bronchodilators (LABA and/or LAMA) ≥ ICS.
  6. ≥ 1 Systemic steroid and/or antibiotic treated exacerbation in the past one year.
  7. Eosinophilic (n=20, blood eosinophils ≥0.200x109/L) and non-eosinophilic (n=20, blood eosinophils <0.200x109/L) phenotypes.
* Healthy controls (n=20)

  1. Asymptomatic
  2. Non-smoking (<10 packyears, quit >6 months)
  3. Normal spirometry (FEV1, FVC, FEV1/FVC ratio: all >LLN)
  4. FeNO < 25 ppb
  5. Non-atopic based on skin-prick test
  6. Negative mannitol provocation test
  7. Younger (n=10, 18-45 years) and older (n=10, >45-75 years) subjects.

Exclusion Criteria:

* Any of the following would exclude the subject from participation in the study:

  1. Previous medical history or evidence of an uncontrolled intercurrent illness that in the opinion of the investigator may compromise the safety of the subject in the study or interfere with evaluation of the investigational product or reduce the subject's ability to participate in the study. Subjects with well-controlled comorbid disease (e.g., hypertension, hyperlipidemia, gastroesophageal reflux disease) on a stable treatment regimen for 15 days prior to Visit 1 are eligible.
  2. Any concomitant respiratory disease that in the opinion of the investigator and/or medical monitor will interfere with the evaluation of the investigational product or interpretation of subject safety or study results (e.g., cystic fibrosis, pulmonary fibrosis, moderate-severe bronchiectasis, allergic bronchopulmonary aspergillosis, Churg-Strauss syndrome, active tuberculosis). In addition for the different groups the following:

     1. Patient with asthma: concomitant COPD.
     2. Patients with COPD: concomitant asthma (former and current)
     3. Healthy subjects: COPD and asthma.
  3. Any clinically relevant abnormal findings in hematology or clinical chemistry (laboratory results from Visit 1), physical examination, vital signs during the screening, which in the opinion of the investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to participate in the study.
  4. Evidence of active liver disease, including jaundice or aspartate transaminase, alanine transaminase, or alkaline phosphatase >1.5 times the upper limit of normal (laboratory results from Visit 1).
  5. GFR <30 ml/min.
  6. Acute upper or lower respiratory infections requiring antibiotics or antiviral medications within 2 weeks prior to Visit 1, during the run-in period, or at Visit 2 (randomization).
  7. A positive human immunodeficiency virus (HIV) test at screening or subject taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
  8. History of sensitivity to any component of the investigational product formulation or a history of drug or other allergy that, in the opinion of the investigator or medical monitor contraindicates their participation.
  9. History of any known primary immunodeficiency disorder excluding asymptomatic selective immunoglobulin A or IgG subclass deficiency.
  10. Receipt of any of the following within 30 days prior to Visit 1:

      1. Immunoglobulin or blood products, or
      2. Receipt of any investigational non-biologic agent within 30 days or 5 half-lives prior Visit 1, whichever is longer.
  11. Pregnant, breastfeeding or lactating females
  12. History of chronic alcohol or drug abuse within 12 months prior to Visit 1.
  13. Planned surgical procedures requiring general anesthesia or in-patient status for > 1 day during the conduct of the study.
  14. Unwillingness or inability to follow the procedures outlined in the protocol.
  15. Concurrent enrollment in another clinical study involving an investigational treatment.
  16. Receipt of any live or attenuated vaccines within 15 days prior to Visit 1.
  17. Long QTc interval on ECG (QTc >480msec).
  18. History of the following cardiac comorbidities:

      1. Life-threatening arrhythmias
      2. Myocardial infarction (NSTEMI or STEMI) less than 6 months before start of the study
      3. Unstable angina
      4. History of severe heart failure
  19. Documented severe hypokalemia (K <3.0 mmol/L) or hypomagnesemia (Mg <0.5 mmol/L).
  20. Life expectancy <6 months.
  21. Hearing impairment.
  22. Oxygen saturation <92% at room air, patients on LTOT, history of chronic respiratory failure (hypercapnia).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
IFN-beta gene and/or protein expression | 12 weeks
  To investigate the potential change in viral induced interferon response in HBECs from baseline and after 12 weeks of treatment with low dose azithromycin or placebo, after stimulation with viral infection mimics (RV16 or Poly (I:C)
Viral load | 12 weeks
  To investigate the potential change in viral load response in HBECs from baseline and 12 weeks of treatment with low dose azithromycin or placebo, after stimulation with viral infection mimics (RV16 or Poly (I:C)

SECONDARY OUTCOMES:
INF-beta gene and/or protein expression | 12 weeks
  To investigate the potential change in viral induced interferon response in HBECs from baseline and after 12 weeks of treatment with low dose azithromycin or placebo, after stimulation with a combination of: viral infection mimics (RV16 or Poly (I:C) +/- allergens (e.g. HDM), +/- scratching of epithelium, +/- smoke exposure.
IL-33 | 12 weeks
  To investigate the potential change in IL-33 response in HBECs from baseline and after 12 weeks of treatment with low dose azithromycin or placebo, after stimulation with viral infection mimics (RV16 or Poly (I:C) in eosinophilic (blood eosinophils >0.2x109/L) and non-eosinophilic (blood eosinophils <0.2x109/L) patients with asthma and COPD.
TSLP | 12 weeks
  To investigate the potential change in IL-33 response in HBECs from baseline and after 12 weeks of treatment with low dose azithromycin or placebo, after stimulation with viral infection mimics (RV16 or Poly (I:C) in eosinophilic (blood eosinophils >0.2x109/L) and non-eosinophilic (blood eosinophils <0.2x109/L) patients with asthma and COPD.
Mast cells, eosinophils, Neutrophils | 12 weeks
  To evaluate the potential change in histologic phenotypes in bronchial biopsies from baseline and after 12 weeks of treatment with low dose azithromycin.
Lung microbiome | 12 weeks
  To evaluate the potential changes in microbiome abundance in BAL-fluid from baseline and after 12 weeks of treatment with low dose azithromycin measured by 16S gene sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Porsbjerg, MD, PhD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg; Therese S Lapperre, MD, PhD, Study Director — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- University Hospital Bispebjerg and Frederiksberg, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No